CLINICAL TRIAL: NCT04751188
Title: Safety and Efficacy of Bezafibrate Plus Ursodesoxicolic Acid in Patients With Primary Biliary Cholangitis Without Response
Brief Title: A Study to Assess Efficacy and Safety of Bezafibrate in Patients With Primary Biliary Cholangitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Jocelyn Serrano Casas, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-2020-2101-031
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Primary Biliary Cirrhosis
Keywords: ursodeoxycholic acid; Bezafibrate
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Bezafibrate; Tablets; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bezafibrate and Ursodeoxycholic acid (Experimental): Bezafibrate 200 mg every 12 hours and ursodeoxycholic acid at a dose of 13 to 15 mg per Kg per day, for 6 months.
  Interventions: Drug: Bezafibrate 200 MG Oral Tablet; Drug: Ursodeoxycholic Acid
- Placebo and Ursodeoxycholic acid (Placebo Comparator): Placebo tablet every 12 hours and ursodeoxycholic acid at a dose of 13 to 15 mg per Kg per day, for 6 months.
  Interventions: Drug: Placebo; Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Bezafibrate 200 MG Oral Tablet — Bezafibrate one tablet every 12 hours for six months.
  Arms: Bezafibrate and Ursodeoxycholic acid
Drug: Placebo — Placebo one tablet every 12 hours for six months.
  Arms: Placebo and Ursodeoxycholic acid
Drug: Ursodeoxycholic Acid — At a dose of 13 to 15 mg per Kg per day.

SUMMARY:
Up to 40% of patients with PBC have an inadequate response to standard treatment with Ursodeoxycholic Acid (UDCA), those patients represent the group in need for additional therapies, having increased risk of disease progression and decreased survival free of liver transplantation.

The main objective of the study is to evaluate safety and efficacy of bezafibrate plus ursodesoxicolic acid in patients with PBC and inadequate response to UDCA.

ELIGIBILITY:
Inclusion Criteria:

* PBC diagnosis (consistent with American Association for the Study of Liver Disease [AASLD]:

  * History of elevated alkaline phosphatase levels.
  * Anti-mitochondrial antibodies positivity
  * Histopathologic evidence of nonsuppurative cholangitis and destruction of small or medium- sized bile ducts.
* Use of ursodeoxycholic acid (UDCA) for at least 12 months at enrollment at a therapeutic dose (13 to 15 mg per Kg per day).
* Evidence of a suboptimal biochemical response to UDCA, defined by the presence of one of the Paris II criteria.
* Written informed consent.
* Age ≥ 18 years.

Exclusion Criteria:

* Hepatic decompensation (ascitis, variceal upper gastrointestinal bleeding, hepatic encephalopathy).
* Coexistence autoimmune hepatitis.
* Bilirrubin >3mg/dl.
* For females, pregnancy or breast-feeding.
* Hepatocellular carcinoma.
* History or presence of spontaneous bacterial peritonitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Biochemical response | 6 months
  Biochemical response is defined as the reduction of alkaline phosphatase lower than 1.5 times the upper normal limit, reduction of aspartate transaminase lower than 1.5 times the upper normal limit and bilirubin lower than 1 mg/dl.

SECONDARY OUTCOMES:
Quality of life | Baseline and 6 months later
  Evaluation of quality of life with the Primary Biliary Cholangitis 40 questionnaire
Pruritus intensity | Baseline and 6 months later
  Evaluation made by the use of visual analogue scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano de Seguro Social, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No